CLINICAL TRIAL: NCT01902498
Title: Multiple Daily Doses of Aspirin to Overcome Hyporesponsiveness Post Cardiac Bypass Surgery (ASACABG)- Part B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Jeremy Paikin, Principal Investigator, Hamilton Health Sciences Corporation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIF-13324
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Postoperative Dysfunction Following Cardiac Surgery
Keywords: aspirin
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aspirin 162mg twice daily (Experimental): Patients will receive 162mg twice daily during the postoperative period, until day 7 postop or the end of hospitalization.
  Interventions: Drug: Aspirin
- Aspirin 325mg daily (Active Comparator): Patients will receive 325mg daily during the postoperative period, until day 7 postop or the end of hospitalization.
  Interventions: Drug: Aspirin
- Aspirin 81mg daily (Active Comparator): Patients will receive 81mg daily during the postoperative period, until day 7 postop or the end of hospitalization.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — Aspirin 81mg po daily x 7days or end of hospitalization. First dose administered on post op day 1.
  Arms: Aspirin 162mg twice daily
Drug: Aspirin — Aspirin 325mg po daily x 7days or end of hospitalization. First dose administered on post op day 1.
  Arms: Aspirin 325mg daily
Drug: Aspirin — Aspirin 162mg po twice daily x 7days or end of hospitalization. First dose administered on post op day 1.
  Arms: Aspirin 81mg daily

SUMMARY:
Cardiac bypass surgery is an important treatment for patients with severely blocked arteries (tubes that delivery oxygen and nutrients to the heart). Hundreds of thousands of these operations are done each year to help relieve patients' chest pain and to prevent future heart attacks. The surgery is done by "bypassing" blood flow around badly clogged arteries by sewing on healthy vessels from another part of the body (usually from the leg or the chest). Aspirin (a blood thinner) is given to patients once a day after their surgery because it stops "sticky" cells in the blood (platelets) from blocking these new vessels (which may lead to a future heart attack).

Research has shown that aspirin does not work as well in people after they have bypass surgery as the investigators might expect (for reasons that are not fully understood). One reason aspirin may not work as well after surgery is because the body makes many more platelets after surgery than it would under normal circumstances. All of these new platelets overwhelm the aspirin and continue to be "sticky" and ready to block off arteries. The investigators believe that giving multiple daily doses of aspirin following bypass surgery is more effective at blocking platelet activity than giving aspirin once daily.

DETAILED DESCRIPTION:
Background:

Cardiovascular disease caused by athero-thrombosis is the number one cause of long-term morbidity and death worldwide. Many patients with advanced coronary disease benefit from Coronary Artery Bypass Graft (CABG) by improving symptoms and increasing their longevity.

However, the benefits of CABG surgery are attenuated by early graft failure. The administration of aspirin in the post-operative period has been shown in randomized controlled trials (RCT) to reduce the risk of graft occlusion, although rates remain unacceptably high. Patients undergoing CABG surgery transiently develop aspirin resistance, which likely contributes to vein graft failure.

The investigators believe the aspirin resistance is a consequence of rapid platelet turnover in the early postoperative period, resulting in a large number of platelets unexposed to aspirin (due to its short half life). The investigators hypothesize that by increasing the frequency of aspirin dosing, the investigators can reverse the aspirin resistance encountered post CABG surgery. The investigators are proposing a RCT comparing two different doses of aspirin (81mg and 325mg daily) to 162mg BID to determine whether multiple daily dosing can overcome aspirin resistance.

(1)Given that platelet production is increased many-fold after CABG surgery (and the short half-life of aspirin), the investigators hypothesize that increasing the frequency of aspirin dosing will lead to the acetylation of a greater number of platelets over the course of the day leading to an improved antiplatelet effect (as measured by serum thromboxane and platelet aggregation assays); (2) The investigators will examine three platelet-related single nucleotide polymorphisms (SNP) that have been implicated in aspirin hyporesponsiveness.

The investigators are proposing a single centre, randomized, open-label, RCT in 60 patients undergoing elective or urgent CABG surgery, to receive ASA 81mg daily, 325mg daily or 162mg bid starting day 1 post-operatively. All patients will receive 325mg 6hrs following the procedure (day of operation) as long as there is no contraindication for antiplatelet therapy (ie significant bleeding) - as per the investigators centre's standard clinical practice. Further details on aspirin administration and outcome measurements are reported below.

ELIGIBILITY:
Inclusion Criteria:

Adult subjects who undergo elective or urgent CABG surgery who are on or off aspirin during the preoperative period with or without valve replacement

Exclusion Criteria:

1. initial platelet count <100,000
2. receiving NSAIDs or other drugs that might interfere with aspirin's platelet-inhibitory effect
3. clinically important bleeding (chest tube drainage >200ml/hr for 6hrs), or bleeding disorders that preclude the use of randomized therapies
4. patients who do not provide informed written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Serum Thromboxane Concentration (ng/ml) | Postoperative Day 4

SECONDARY OUTCOMES:
Arachidonic Acid Induced Light Transmission Aggregometry (LTA): Aggregation will be expressed as the maximum percent change in light transmittance from baseline, with platelet-poor plasma used as a reference. | Postoperative Day 4
DNA genetic analyses for single nucleotide polymorphisms | A single preoperative blood sample was drawn (on average 1 day prior to surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Paikin, MD, Principal Investigator — Cardiology Fellow; John Eikelboom, MBBS, Principal Investigator — Hematologist, PHRI researcher; Richard Whitlock, MD, Principal Investigator — Cardiac Surgeon, PHRI researcher; Guillaume Pare, MD, Principal Investigator — Medical Biochemist, PHRI researcher; Jack Hirsh, MD, Principal Investigator — Hematologist, Professor Emeritus, PHRI researcher
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada